CLINICAL TRIAL: NCT06957444
Title: Rate of Allergic Contact Dermatitis and Cosmetic Outcomes for Three Wound Closure Techniques in Joint Arthroplasty Patients: A Randomized, Controlled Trial
Brief Title: Rate of Allergic Contact Dermatitis and Cosmetic Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Benjamin Frye, Associate Professor, Fellowship Director Adult Reconstruction, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2503134113
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Allergic Contact Dermatitis; Osteoarthritis, Hip; Osteoarthritis, Knee
MeSH Terms: conditions — Dermatitis, Allergic Contact; Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sylke Adhesive Dressing (Active Comparator): Topical Wound Closure to be applied once the deep wound closure is secured after Total Knee or Total Hip Arthroplasty
  Interventions: Procedure: Sylke Adhesive Dressing
- Exofin Skin Glue (Active Comparator): Topical Wound Closure to be applied once the deep wound closure is secured after Total Knee or Total Hip Arthroplasty
  Interventions: Procedure: Exofin Skin Glue
- Suture Strip Plus (Active Comparator): Topical Wound Closure to be applied once the deep wound closure is secured after Total Knee or Total Hip Arthroplasty
  Interventions: Procedure: Suture Strip Plus

INTERVENTIONS:
Procedure: Sylke Adhesive Dressing — Topical wound closure device, made from silk fibroin woven mesh coated with a pressure-sensitive acrylic adhesive.
  Arms: Sylke Adhesive Dressing
Procedure: Exofin Skin Glue — 2-octil cyanoacrylate formulation, applied using a soft and flexible applicator.
  Arms: Exofin Skin Glue
Procedure: Suture Strip Plus — Flexible wound closure strip designed for primary wound closure made up of macroporous non-woven polyamide with a pressure sensitive adhesive.
  Arms: Suture Strip Plus

SUMMARY:
The patients from the Department of Orthopaedics Center for Joint Replacement will be asked to participate in the study. These patients will be randomized to one of three wound closure products, Sylke adhesive dressing, Exofin skin glue, or Suture Strip Plus. Participants will be asked to take a photograph of the incision 4 days after surgery to submit via MyChart for review by the WVU Department of Dermatology Team. All patients will be evaluated at their regular 2-week, 6-week, and 3-month post-operative visits where clinical photographs will be submitted for independent review by the WVU Department of Dermatology Team to assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign the informed consent
* Patients presenting to the WVU Medicine Center for Joint Replacement who have a primary TKA or THA surgery scheduled
* Patients with surgical wounds closed by 2-0 vicryl and barbed, running v-loc suture (assessed in OR)
* Active MyChart account and the ability to take and upload a photo in that system

Exclusion Criteria:

* Patients scheduled for a revision THA or revision TKA
* THA used for treatment of a fracture
* Patients participating in other studies that might have involve medications such as antibiotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Rate of allergic contact dermatitis (4 Days Post Op) | 4 Days Post-Op
  Percentage of participants exhibiting allergic contact dermatitis as determined by using the International Contact Dermatitis Research Group (ICDRG) scale with any reaction including and above "Weak Positive" being included in this rate of allergic contact dermatitis:
  Negative (0): No reaction. Doubtful (+?): Slight erythema (redness) without infiltration. Weak positive (+): Erythema, infiltration, possibly papules. Strong positive (++): Erythema, infiltration, papules, vesicles. Extreme positive (+++): Intense erythema, infiltration, coalescing vesicles, bullous reaction.
Rate of allergic contact dermatitis (2 Weeks Post Op) | 2 Weeks Post-Op
  Percentage of participants exhibiting allergic contact dermatitis as determined by using the International Contact Dermatitis Research Group (ICDRG) scale with any reaction including and above "Weak Positive" being included in this rate of allergic contact dermatitis:
  Negative (0): No reaction. Doubtful (+?): Slight erythema (redness) without infiltration. Weak positive (+): Erythema, infiltration, possibly papules. Strong positive (++): Erythema, infiltration, papules, vesicles. Extreme positive (+++): Intense erythema, infiltration, coalescing vesicles, bullous reaction.
Rate of allergic contact dermatitis (6 Weeks Post Op) | 6 Weeks Post-Op
  Percentage of participants exhibiting allergic contact dermatitis as determined by using the International Contact Dermatitis Research Group (ICDRG) scale with any reaction including and above "Weak Positive" being included in this rate of allergic contact dermatitis:
  Negative (0): No reaction. Doubtful (+?): Slight erythema (redness) without infiltration. Weak positive (+): Erythema, infiltration, possibly papules. Strong positive (++): Erythema, infiltration, papules, vesicles. Extreme positive (+++): Intense erythema, infiltration, coalescing vesicles, bullous reaction.
Rate of allergic contact dermatitis (3 Months Post Op) | 3 Months Post-Op
  Percentage of participants exhibiting allergic contact dermatitis as determined by using the International Contact Dermatitis Research Group (ICDRG) scale with any reaction including and above "Weak Positive" being included in this rate of allergic contact dermatitis:
  Negative (0): No reaction. Doubtful (+?): Slight erythema (redness) without infiltration. Weak positive (+): Erythema, infiltration, possibly papules. Strong positive (++): Erythema, infiltration, papules, vesicles. Extreme positive (+++): Intense erythema, infiltration, coalescing vesicles, bullous reaction.

SECONDARY OUTCOMES:
Difference in Cosmetic Outcome (4 Days Post-Op) | 4 Days Post-Op
  The Scar Cosmesis Assessment and Rating (SCAR) scale is a validated tool used to assess the quality of postoperative scars. The SCAR scale measures postoperative scar cosmesis with scores ranging from 0 (best possible scar) to 15 (worst possible scar). The assessment includes both clinician and patient items, ensuring a comprehensive evaluation.
Difference in Cosmetic Outcome (2 Weeks Post-Op) | 2 Weeks Post-Op
  The Scar Cosmesis Assessment and Rating (SCAR) scale is a validated tool used to assess the quality of postoperative scars. The SCAR scale measures postoperative scar cosmesis with scores ranging from 0 (best possible scar) to 15 (worst possible scar). The assessment includes both clinician and patient items, ensuring a comprehensive evaluation.
Difference in Cosmetic Outcome (6 Weeks Post-Op) | 6 Weeks Post-Op
  The Scar Cosmesis Assessment and Rating (SCAR) scale is a validated tool used to assess the quality of postoperative scars. The SCAR scale measures postoperative scar cosmesis with scores ranging from 0 (best possible scar) to 15 (worst possible scar). The assessment includes both clinician and patient items, ensuring a comprehensive evaluation.
Difference in Cosmetic Outcome (3 Months Post-Op) | 3 Months Post-Op
  The Scar Cosmesis Assessment and Rating (SCAR) scale is a validated tool used to assess the quality of postoperative scars. The SCAR scale measures postoperative scar cosmesis with scores ranging from 0 (best possible scar) to 15 (worst possible scar). The assessment includes both clinician and patient items, ensuring a comprehensive evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Frye, MD, Principal Investigator — West Virginia University Department of Orthopaedics
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao E, Tarkin IS, Moloney GB. Subcuticular Barbed Suture and Skin Glue Wound Closure Decreases Reoperation and Length of Stay in Geriatric Hip Fractures When Compared With Staples. J Am Acad Orthop Surg Glob Res Rev. 2021 Oct 4;5(10):e21.00205. doi: 10.5435/JAAOSGlobal-D-21-00205. PMID 34605793
- [Background] Ali E, Makhdom AM. Association of Surgical Adhesive and Glue System With Incidence of Allergic Dermatitis Post Unilateral and Staged Bilateral Total Knee Arthroplasty. Cureus. 2024 Apr 23;16(4):e58827. doi: 10.7759/cureus.58827. eCollection 2024 Apr. PMID 38654960
- [Background] Ricciardo BM, Nixon RL, Tam MM, Radic RR, Ricciardo BJ. Allergic Contact Dermatitis to Dermabond Prineo After Elective Orthopedic Surgery. Orthopedics. 2020 Nov 1;43(6):e515-e522. doi: 10.3928/01477447-20200827-01. Epub 2020 Sep 3. PMID 32882052
- [Background] Pannu CD, Farooque Md K. Allergic Contact Dermatitis to Octyl Cyanoacrylate Skin Glue After Surgical Wound Closure: A Systematic Review. Dermatitis. 2024 Sep-Oct;35(5):443-466. doi: 10.1089/derm.2023.0342. Epub 2024 Feb 21. PMID 38386590
- [Background] Kim D, Lee NR, Park SY, Jun M, Lee K, Kim S, Park CS, Liu KH, Choi EH. As in Atopic Dermatitis, Nonlesional Skin in Allergic Contact Dermatitis Displays Abnormalities in Barrier Function and Ceramide Content. J Invest Dermatol. 2017 Mar;137(3):748-750. doi: 10.1016/j.jid.2016.10.034. Epub 2016 Nov 5. No abstract available. PMID 27826010
- [Background] Zhang W, Xu J, Qu S, Peng H. The impact of allergic contact dermatitis on the inflammatory response and repair in wound healing process. Front Med (Lausanne). 2025 Feb 19;12:1524198. doi: 10.3389/fmed.2025.1524198. eCollection 2025. PMID 40046929
- [Background] Rouhani DS, Singh NK, Chao JJ, Almutairi A, Seradj MH, Badowski-Platz R, Toranto JD, Mofid MM. Superiority of a Silk Surgical Site Wound Closure Device over Synthetic Dressings. Plast Reconstr Surg. 2024 Dec 1;154(6):1233-1244. doi: 10.1097/PRS.0000000000011316. Epub 2024 Feb 7. PMID 38330504
- [Background] Rouhani DS, Singh NK, Chao JJ, Almutairi A, Badowski-Platz R, Seradj MH, Mofid MM. Silk Bioprotein as a Novel Surgical-Site Wound Dressing: A Prospective, Randomized, Single-Blinded, Superiority Clinical Trial. Aesthet Surg J Open Forum. 2023 Oct 20;5:ojad071. doi: 10.1093/asjof/ojad071. eCollection 2023. PMID 37899912
- [Background] Custis T, Armstrong AW, King TH, Sharon VR, Eisen DB. Effect of Adhesive Strips and Dermal Sutures vs Dermal Sutures Only on Wound Closure: A Randomized Clinical Trial. JAMA Dermatol. 2015 Aug;151(8):862-7. doi: 10.1001/jamadermatol.2015.0174. PMID 25875131
- [Background] Takayama S, Yamamoto T, Tsuchiya C, Noguchi H, Sato J, Ishii Y. Comparing Steri-Strip and surgical staple wound closures after primary total knee arthroplasties. Eur J Orthop Surg Traumatol. 2017 Jan;27(1):113-118. doi: 10.1007/s00590-016-1848-x. Epub 2016 Sep 6. PMID 27600333
- [Background] Johansen JD, Aalto-Korte K, Agner T, Andersen KE, Bircher A, Bruze M, Cannavo A, Gimenez-Arnau A, Goncalo M, Goossens A, John SM, Liden C, Lindberg M, Mahler V, Matura M, Rustemeyer T, Serup J, Spiewak R, Thyssen JP, Vigan M, White IR, Wilkinson M, Uter W. European Society of Contact Dermatitis guideline for diagnostic patch testing - recommendations on best practice. Contact Dermatitis. 2015 Oct;73(4):195-221. doi: 10.1111/cod.12432. Epub 2015 Jul 14. PMID 26179009
- [Background] Kantor J. Reliability and Photographic Equivalency of the Scar Cosmesis Assessment and Rating (SCAR) Scale, an Outcome Measure for Postoperative Scars. JAMA Dermatol. 2017 Jan 1;153(1):55-60. doi: 10.1001/jamadermatol.2016.3757. PMID 27806156